CLINICAL TRIAL: NCT03977025
Title: Evaluation of Alzheimer's Biomarkers in Cerebrospinal Fluid and Peripheral Blood of Elderly Patients Undergoing Surgery in the HCUCH.
Brief Title: Alzheimer Biomarkers on CSF of Elderly Patients Undergoing Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Sergio Vera, Principal Investigator, University of Chile
Other Study IDs: Saval 018
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lumbar punction — Patients will be evaluated prior to surgery with the Montreal Cognitive Assessment (MoCA) to determine the presence of cognitive impairment, and CSF samples, obtained by lumbar punction, will be analyzed by immunodetection of Aβ40, Aβ42, tau and ptau with multiplex technology
  Other Names: Montreal Cognitive Assessment

SUMMARY:
Dementia is a syndrome characterized by cognitive and behavioral impairment in older adults, which usually manifests as memory loss, communication difficulties or changes in mood. Dementias affect around 50 million people in the world, having an impact on their ability to carry out their daily activities, often requiring family and social support.

The main cause of dementia in Chile and in the world is Alzheimer's disease (AD), which is characterized by affecting large areas of the cerebral cortex and hippocampus, manifesting mainly in alterations in selective memory. The pathogenesis of AD involves the neuronal accumulation of β-amyloid (Aβ) proteins in the form of extracellular plaques, and tau, which gives rise to neurofibrillary tangles. AD diagnosis is usually made based on clinical criteria, however, the accurate diagnosis of AD is clinical-neuropathological. Several studies have supported the neuropathological study based on the presence of Aβ and tau proteins in cerebrospinal fluid (CSF), using them as biomarkers of the disease, which has allowed updating the definition of AD based on them. However, our country does not perform a study of dementia biomarkers in CSF, which is essential for the diagnosis of certainty of the pathology.

The objective of this project is to evaluate a set of biomarkers of EA (tau, ptau, Aβ) in CSF and blood of elderly patients who will undergo surgery in the Clinical Hospital of the University of Chile (HCUCH) and in whom it is performed lumbar puncture (LP) by anesthesia, to detect those patients who have these CSF biomarkers and who show lower performance in cognitive evaluations. For this, it is intended to mount a biobank of CSF samples with samples of 30 subjects by conducting a clinical pilot study. Patients will be evaluated prior to surgery with the Montreal Cognitive Assessment (MoCA) to determine the presence of cognitive impairment, and CSF samples, obtained by LP, will be analyzed by immunodetection of Aβ40, Aβ42, tau and ptau with multiplex technology. In addition, tau will be detected in platelets by Western Blot of blood samples from patients, and the relationship between plateau tau levels and biomarkers in CSF will be evaluated. Finally, the correlation between performance in cognitive assessment and levels of biomarkers in blood and CSF will be evaluated, in order to assess the usefulness of these markers in the detection of the presence of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 65 years who will undergo surgery in the HCUCH (for any reason) and who require lumbar puncture for anesthesia.
* Autovalent, with no history of dementia, with MoCA ≥ 20 points (score adapted to the Chilean population).
* The subjects will not be carriers of medical, neurological or psychiatric pathologies that could affect their participation in the study or its results. The presence of chronic pathologies will be admitted, as long as they are under stable treatment and without evidence of decompensation in the last 3 months.

Exclusion Criteria:

* Antecedents of being carriers of dementia or symptomatic neurodegenerative disease.
* Medical or surgical decompensated pathology.
* Contraindication of lumbar puncture.
* Physical or mental inability to consent to study entry.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients who will undergo surgery in the HCUCH, for any reason
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 1 day
  Correlate the degree of cognitive deterioration obtained in the MOCA evaluation with the levels of biomarkers in CSF and blood.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Vera, MD, Principal Investigator — University of Chile
Locations (1):
- University of Chile Clinical Hospital, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), American Psychiatric Association. 2013.
- [Background] Scheltens P, Blennow K, Breteler MM, de Strooper B, Frisoni GB, Salloway S, Van der Flier WM. Alzheimer's disease. Lancet. 2016 Jul 30;388(10043):505-17. doi: 10.1016/S0140-6736(15)01124-1. Epub 2016 Feb 24. PMID 26921134
- [Background] Wang J, Gu BJ, Masters CL, Wang YJ. A systemic view of Alzheimer disease - insights from amyloid-beta metabolism beyond the brain. Nat Rev Neurol. 2017 Sep 29;13(10):612-623. doi: 10.1038/nrneurol.2017.111. PMID 28960209
- [Background] Masters CL, Bateman R, Blennow K, Rowe CC, Sperling RA, Cummings JL. Alzheimer's disease. Nat Rev Dis Primers. 2015 Oct 15;1:15056. doi: 10.1038/nrdp.2015.56. PMID 27188934
- [Background] Alzheimer's Disease International publication team. From plan to impact. Progress towards targets of the Global action plan on dementia. Alzheimer's Disease International. 2018.
- [Background] Parra MA, Baez S, Allegri R, Nitrini R, Lopera F, Slachevsky A, Custodio N, Lira D, Piguet O, Kumfor F, Huepe D, Cogram P, Bak T, Manes F, Ibanez A. Dementia in Latin America: Assessing the present and envisioning the future. Neurology. 2018 Jan 30;90(5):222-231. doi: 10.1212/WNL.0000000000004897. Epub 2018 Jan 5. PMID 29305437
- [Background] Fuentes P, Albala C. An update on aging and dementia in Chile. Dement Neuropsychol. 2014 Oct-Dec;8(4):317-322. doi: 10.1590/S1980-57642014DN84000003. PMID 29213920
- [Background] Gremer L, Scholzel D, Schenk C, Reinartz E, Labahn J, Ravelli RBG, Tusche M, Lopez-Iglesias C, Hoyer W, Heise H, Willbold D, Schroder GF. Fibril structure of amyloid-beta(1-42) by cryo-electron microscopy. Science. 2017 Oct 6;358(6359):116-119. doi: 10.1126/science.aao2825. Epub 2017 Sep 7. PMID 28882996
- [Background] DeVos SL, Miller RL, Schoch KM, Holmes BB, Kebodeaux CS, Wegener AJ, Chen G, Shen T, Tran H, Nichols B, Zanardi TA, Kordasiewicz HB, Swayze EE, Bennett CF, Diamond MI, Miller TM. Tau reduction prevents neuronal loss and reverses pathological tau deposition and seeding in mice with tauopathy. Sci Transl Med. 2017 Jan 25;9(374):eaag0481. doi: 10.1126/scitranslmed.aag0481. PMID 28123067
- [Background] Ittner A, Chua SW, Bertz J, Volkerling A, van der Hoven J, Gladbach A, Przybyla M, Bi M, van Hummel A, Stevens CH, Ippati S, Suh LS, Macmillan A, Sutherland G, Kril JJ, Silva AP, Mackay JP, Poljak A, Delerue F, Ke YD, Ittner LM. Site-specific phosphorylation of tau inhibits amyloid-beta toxicity in Alzheimer's mice. Science. 2016 Nov 18;354(6314):904-908. doi: 10.1126/science.aah6205. PMID 27856911
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Buerger K, Ewers M, Pirttila T, Zinkowski R, Alafuzoff I, Teipel SJ, DeBernardis J, Kerkman D, McCulloch C, Soininen H, Hampel H. CSF phosphorylated tau protein correlates with neocortical neurofibrillary pathology in Alzheimer's disease. Brain. 2006 Nov;129(Pt 11):3035-41. doi: 10.1093/brain/awl269. Epub 2006 Sep 29. PMID 17012293
- [Background] Mattsson N, Zetterberg H, Hansson O, Andreasen N, Parnetti L, Jonsson M, Herukka SK, van der Flier WM, Blankenstein MA, Ewers M, Rich K, Kaiser E, Verbeek M, Tsolaki M, Mulugeta E, Rosen E, Aarsland D, Visser PJ, Schroder J, Marcusson J, de Leon M, Hampel H, Scheltens P, Pirttila T, Wallin A, Jonhagen ME, Minthon L, Winblad B, Blennow K. CSF biomarkers and incipient Alzheimer disease in patients with mild cognitive impairment. JAMA. 2009 Jul 22;302(4):385-93. doi: 10.1001/jama.2009.1064. PMID 19622817
- [Background] Clark CM, Pontecorvo MJ, Beach TG, Bedell BJ, Coleman RE, Doraiswamy PM, Fleisher AS, Reiman EM, Sabbagh MN, Sadowsky CH, Schneider JA, Arora A, Carpenter AP, Flitter ML, Joshi AD, Krautkramer MJ, Lu M, Mintun MA, Skovronsky DM; AV-45-A16 Study Group. Cerebral PET with florbetapir compared with neuropathology at autopsy for detection of neuritic amyloid-beta plaques: a prospective cohort study. Lancet Neurol. 2012 Aug;11(8):669-78. doi: 10.1016/S1474-4422(12)70142-4. Epub 2012 Jun 28. Erratum In: Lancet Neurol. 2012 Aug;11(8):658. PMID 22749065
- [Background] Clark CM, Schneider JA, Bedell BJ, Beach TG, Bilker WB, Mintun MA, Pontecorvo MJ, Hefti F, Carpenter AP, Flitter ML, Krautkramer MJ, Kung HF, Coleman RE, Doraiswamy PM, Fleisher AS, Sabbagh MN, Sadowsky CH, Reiman EP, Zehntner SP, Skovronsky DM; AV45-A07 Study Group. Use of florbetapir-PET for imaging beta-amyloid pathology. JAMA. 2011 Jan 19;305(3):275-83. doi: 10.1001/jama.2010.2008. PMID 21245183
- [Background] Seo SW, Ayakta N, Grinberg LT, Villeneuve S, Lehmann M, Reed B, DeCarli C, Miller BL, Rosen HJ, Boxer AL, O'Neil JP, Jin LW, Seeley WW, Jagust WJ, Rabinovici GD. Regional correlations between [11C]PIB PET and post-mortem burden of amyloid-beta pathology in a diverse neuropathological cohort. Neuroimage Clin. 2016 Nov 11;13:130-137. doi: 10.1016/j.nicl.2016.11.008. eCollection 2017. PMID 27981028
- [Background] Blennow K, Zetterberg H. Biomarkers for Alzheimer's disease: current status and prospects for the future. J Intern Med. 2018 Dec;284(6):643-663. doi: 10.1111/joim.12816. Epub 2018 Aug 19. PMID 30051512
- [Background] Slachevsky A, Guzman-Martinez L, Delgado C, Reyes P, Farias GA, Munoz-Neira C, Bravo E, Farias M, Flores P, Garrido C, Becker JT, Lopez OL, Maccioni RB. Tau Platelets Correlate with Regional Brain Atrophy in Patients with Alzheimer's Disease. J Alzheimers Dis. 2017;55(4):1595-1603. doi: 10.3233/JAD-160652. PMID 27911301
- [Background] Farias G, Perez P, Slachevsky A, Maccioni RB. Platelet tau pattern correlates with cognitive status in Alzheimer's disease. J Alzheimers Dis. 2012;31(1):65-9. doi: 10.3233/JAD-2012-120304. PMID 22495344
- [Background] Kern S, Zetterberg H, Kern J, Zettergren A, Waern M, Hoglund K, Andreasson U, Wetterberg H, Borjesson-Hanson A, Blennow K, Skoog I. Prevalence of preclinical Alzheimer disease: Comparison of current classification systems. Neurology. 2018 May 8;90(19):e1682-e1691. doi: 10.1212/WNL.0000000000005476. Epub 2018 Apr 13. PMID 29653987
- [Background] Delgado C, Araneda A, Behrens MI. Validation of the Spanish-language version of the Montreal Cognitive Assessment test in adults older than 60 years. Neurologia (Engl Ed). 2019 Jul-Aug;34(6):376-385. doi: 10.1016/j.nrl.2017.01.013. Epub 2017 Mar 30. English, Spanish. PMID 28364958